CLINICAL TRIAL: NCT04123080
Title: A Novel Technique Using Endoscopic Band Ligation for Removal of Long-stalked (>10 mm) Pedunculated Colon Polyps
Brief Title: A Technique Using EBL for Removal of Pedunculated Colon Polyps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uijeongbu St. Mary Hospital (Other)
Responsible Party: Principal Investigator, Hiun Suk Chae, Professor, Uijeongbu St. Mary Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UC12RISI0173
Record Dates: First submitted 2019-10-07; First posted 2019-10-10 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Colonic Polyp
Keywords: Colonic Polyp; Endoscopic mucosal resection
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EBL group (Experimental): Removal of large long-stalked pedunculated colonic polyps using band ligations
  Interventions: Device: Endoscopic band ligation assisted polypectomy

INTERVENTIONS:
Device: Endoscopic band ligation assisted polypectomy — A conventional upper endoscope loaded with a band ligator was inserted in the colon and was advanced to the site of the pedunculated polyp. After approaching the lateral side of the stalk and grasping the mid-portion of the stalk using a tripod grasper. Then, the rubber band was released from the cap to ligate the stalk. Thereafter, we performed polypectomy of the remaining stalk just above the ligation by extending the electrosurgical snare.

SUMMARY:
Bleeding is the most common complication associated with polypectomy of large pedunculated colonic polyp. Although several techniques have been developed to minimize bleeding, none of these methods has become the gold standard. To prevent post-polypectomy bleeding effectively, the investigators developed and attempted a new endoscopic technique for removal of large long-stalked pedunculated colonic polyps using band ligations. This study aims to evaluate the safety and efficacy of a novel technique using endoscopic band ligation for removal of long-stalked pedunculated colon polyps.

DETAILED DESCRIPTION:
A prospective single-center study was conducted. Targeted polyps were large (head size >10 mm) with long stalk length (>10 mm) in the distal colon. After finding target lesions by standard colonoscopy, conventional upper endoscopy with rubber band (endoscopic band ligation, EBL) was applied to squeeze the mid-portion of the stalk to form an omega shape, which had the dual effect of ligation and compression of feeding blood vessels. After strangulation of the stalk, snare polypectomy was performed at the stalk site just above the ligation. The investigators evaluated several parameters, including completeness of resection, procedure time, and complications, including immediate postpolypectomy bleeding, delayed postpolypectomy bleeding, and perforation.

ELIGIBILITY:
Inclusion Criteria:

* Polyps with head >10 mm and stalk length >10 mm;
* Location at the distal segments of the colon; and
* Benign features under endoscopic inspection (absence of ulceration and induration or friability).

Exclusion Criteria:

* Patients who refuse to sign the consent

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-04-01 (Actual); Primary Completion 2014-01-31 (Actual); Study Completion 2014-01-31 (Actual)

PRIMARY OUTCOMES:
Rate of completed polyp resection | Immediately after the intervention
  a lesion-free margin with both the lateral and basal tissues free of pathology
Procedure time | during the procedure
  From approaching the the stalk to snare polypectomy with electrosurgical snare
Rate of immediate postpolypectomy bleeding | during the procedure
  pulsating bleeding or oozing lasting more than 60 s immediately after polypectomy or requiring endoscopic intervention.
Rate of delayed postpolypectomy bleeding | 30 days after procedure
  gross rectal bleeding, bleeding requiring endoscopic or radiological hemostasis, or transfusions requiring surgery
Rate of perforation | 30 days after procedure
  endoscopically observed colonic wall penetration, or perforation detected after endoscopy by radiological examination including abdomen CT.

CONTACTS AND LOCATIONS:
Overall Officials: Hiun-Suk Chae, Professor, Principal Investigator — Uijeongbu St. Mary's Hospital, The Catholic University of Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fyock CJ, Draganov PV. Colonoscopic polypectomy and associated techniques. World J Gastroenterol. 2010 Aug 7;16(29):3630-7. doi: 10.3748/wjg.v16.i29.3630. PMID 20677334
- [Background] Ferlitsch M, Moss A, Hassan C, Bhandari P, Dumonceau JM, Paspatis G, Jover R, Langner C, Bronzwaer M, Nalankilli K, Fockens P, Hazzan R, Gralnek IM, Gschwantler M, Waldmann E, Jeschek P, Penz D, Heresbach D, Moons L, Lemmers A, Paraskeva K, Pohl J, Ponchon T, Regula J, Repici A, Rutter MD, Burgess NG, Bourke MJ. Colorectal polypectomy and endoscopic mucosal resection (EMR): European Society of Gastrointestinal Endoscopy (ESGE) Clinical Guideline. Endoscopy. 2017 Mar;49(3):270-297. doi: 10.1055/s-0043-102569. Epub 2017 Feb 17. PMID 28212588
- [Background] Baron TH, Wong Kee Song LM. Endoscopic variceal band ligation. Am J Gastroenterol. 2009 May;104(5):1083-5. doi: 10.1038/ajg.2008.17. No abstract available. PMID 19417747
- [Background] Carmo J, Marques S, Chapim I, Barreiro P, Bispo M, Chagas C. Elastic band ligation for the removal of a colonic tubular adenoma in a diverticulum. Endoscopy. 2015;47 Suppl 1 UCTN:E490-1. doi: 10.1055/s-0034-1393142. Epub 2015 Oct 19. No abstract available. PMID 26479300